CLINICAL TRIAL: NCT06138145
Title: Testing the Impact of Appeals to Diversity and Inclusion in Pediatric Clinical Research Study Enrollment Videos: a Baseline Assessment Study
Brief Title: Inclusion Appeal Videos and Intent to Register for Pediatric Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Kevin Johnson, David L. Cohen University Professor of Pediatrics, Biomedical Informatics, Computer Science and Science Communication, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-019955
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Patient Participation; Pediatric ALL
Keywords: Inclusion Study; African American Study; African American Pediatrics; Appeal Videos
MeSH Terms: conditions — Patient Participation; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): Text introduction from the Registry, with a gift card.
  Interventions: Other: Video; Behavioral: Survey
- Generic (Experimental): Video detailing the Registry's objectives, no tailoring, with a gift card.
  Interventions: Other: Video; Behavioral: Survey
- Appeal (Experimental): Generic video edited to include a tailored appeal, with a gift card.
  Interventions: Other: Video; Behavioral: Survey
- Ink pen (no) Incentive: (Sham Comparator): Similar to control but received a University ink pen.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Other: Video — Different videos were shown for the generic and appeal groups. No videos were shown to the control or ink-pen incentive groups
  Arms: Appeal; Control; Generic
Behavioral: Survey — Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.

SUMMARY:
An informational video about joining a Research Notification Registry is being compared with a version of the video tailored to African/ African American parents, reminding them about the importance of their being included in clinical trials. African/African American parents and caregivers of children under 13 years of age are targeted.

DETAILED DESCRIPTION:
Improving diversity in research projects and national data repositories is critical to providing safe and effective care to marginalized groups. Unfortunately, certain groups such as African Americans are inadequately represented in much of the available data and in current clinical trials. Recently, investigators have begun employing new messaging approaches to increase diversity in clinical trial enrollment. These messages are typically designed to inform, with no appeal for specific groups to act, and no tailoring that takes into account specific groups. Very little is known about the potential impact of inclusion appeals--direct appeals to historically marginalized groups calling on their need to be included in research studies. Applying the science of appeals to recruitment messages may improve the effectiveness of educational videos and lead to greater participation in research. This pilot study proposes to empirically study whether an inclusion appeal increases decisions to enroll children in studies.

ELIGIBILITY:
Inclusion:

1. English speaking
2. Self-identified African or African American
3. Not already enrolled in any research participant registry, no history of clinical trial participation
4. At least one child in their care age newborn to 13

Exclusion:

1. Parents with children over the age of 13
2. Non-English speakers
3. Previously enrolled in Children's Hospital of Philadelphia registry, history of clinical trial participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHOP Primary Care, Cobbs Creek, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Johnson KB, Iannone SL, Furth SL, Taylor L, Tan ASL. Culturally Tailored Messages and Trial Registry Enrollment: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2444229. doi: 10.1001/jamanetworkopen.2024.44229. PMID 39531233
- See also: Inclusion Study References — https://upenn.box.com/s/jmnzb7zdeh70ojwbvntlvkfgdhei6el1

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No Video w/ monetary incentive
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
- Generic: Generic video w/ monetary incentive
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
- Appeal: Appeal video w/ monetary incentive
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
- Ink Pen (no) Incentive: Non-Incentive and no video
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
Period: Overall Study
Arm/Group | Control | Generic | Appeal | Ink Pen (no) Incentive
Started | 29 | 30 | 34 | 32
Completed | 29 | 30 | 33 | 32
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Generic | Appeal | Ink Pen (no) Incentive | Total
Number analyzed (Participants) | 29 | 30 | 34 | 32 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 34 | 32 | 125
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32.3 [20 to 57] | 32.8 [20 to 57] | 32.3 [20 to 57] | 33.1 [20 to 57] | 32.6 [20 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 30 | 28 | 110
  Male | 3 | 4 | 4 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 28 | 28 | 30 | 29 | 115
  White | 1 | 1 | 0 | 2 | 4
  More than one race | 0 | 0 | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 34 | 32 | 125

OUTCOME MEASURES:

1. Primary Outcome: Participants' Decision to Enroll in the CHOP Pediatric Clinical Trials Registry
Description: Number of Participants with who made the decision to enroll in the CHOP pediatric clinical trials registry.
Time Frame: Up to 40 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Ink Pen (no) Incentive: Similar to control but received a University ink pen.
Arm/Group | Control | Generic | Appeal | Ink Pen (no) Incentive
Number analyzed (Participants) | 29 | 30 | 34 | 32
Participants | 29 | 30 | 34 | 32
Statistical Analysis 1: Comparison: Control vs Generic vs Appeal vs Ink Pen (no) Incentive; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Control vs Generic vs Appeal vs Ink Pen (no) Incentive; Test type: Other; p < 0.05, Mann-Whitney U test
Statistical Analysis 3: Comparison: Control vs Generic vs Appeal vs Ink Pen (no) Incentive; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored in this study, as participation concluded immediately upon completion of the survey. This study was classified as low risk, as it involved only the collection of survey responses without any medical interventions, treatments, or procedures. Given the minimal risk associated with survey-based research, ongoing safety monitoring was not required. Participants were informed that they could discontinue the survey at any time if they experienced discomfort.
Description: Adverse events were not monitored in this study, as participation concluded immediately upon completion of the survey. This study was classified as low risk, as it involved only the collection of survey responses without any medical interventions, treatments, or procedures. Given the minimal risk associated with survey-based research, ongoing safety monitoring was not required. Participants were informed that they could discontinue the survey at any time if they experienced discomfort.
Groups:
- Control: Text introduction from the Registry, with a gift card.
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
- Generic: Video detailing the Registry's objectives, no tailoring, with a gift card.
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
- Appeal: Generic video edited to include a tailored appeal, with a gift card.
  Video: Different videos were shown for Arms B and C. No Video was shown for Group A or D.
  Survey: Survey about participant's demographics, information source trust, and clinical trials knowledge. Also includes question about whether the participant is interested in enrolling in the Pediatric Trials Notification System.
Arm/Group | Control | Generic | Appeal | Ink Pen (no) Incentive:
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Several factors may affect the interpretation of this study. The sample was drawn from a few urban sites, which could limit the representation of marginalized groups. The fourth study arm was recruited six months later, potentially influencing baseline trust and timing. Participants knew about the incentive before consenting, which may have shaped trust perceptions. Only baseline self-reported data were collected, with no follow-up to assess changes in trust or knowledge after the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT06138145/Prot_SAP_000.pdf